CLINICAL TRIAL: NCT00739492
Title: Testing Strategies for Weight Loss, II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: William and Flora Hewlett Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01074
Record Dates: First submitted 2008-05-20; First posted 2008-08-21 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
Keywords: weight loss, obesity, financial incentives
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): deposit based incentive
  Interventions: Behavioral: financial incentives
- 2 (Active Comparator): deposit based incentive framed with "maintenance" period
  Interventions: Behavioral: financial incentives
- 3 (No Intervention): Control arm, no financial incentive

INTERVENTIONS:
Behavioral: financial incentives — financial incentives based on attaining weight loss goals
  Arms: 1; 2

SUMMARY:
In the pilot study, Testing Strategies for Weight Loss, we tested two different approaches using financial incentives to encourage weight loss. In the first, we built on previous work showing the effectiveness of 'deposit contracts', in which subjects are given the opportunity to put their own money at risk if they do not lose weight. In this incentive condition, subjects received a direct payment conditional on daily weight loss, and an optional additional payment based on their own contributions to the deposit contract. We matched their contribution 1:1 to make the option of depositing their own money attractive to this predominantly low SES population. In the second approach we built on our own prior work using lotteries to promote drug adherence. In this incentive condition, participants are entered into a daily lottery, and receive any payoffs they earn from the lottery only if they stay on track with their weight-loss goal. Given their popularity in the general population, lotteries hold the promise of providing a cost-effective means of motivating weight loss and making efforts to lose weight more salient to obese patients. Results from this trial indicate significantly higher weight loss in the incentive arms of the trial than in the control group. The low lost to follow-up rates suggest that this approach to providing daily feedback to keep weight loss salient among participants is feasible. Incentive participants who completed the study called in their daily weights an average 95.8% of the time. 17/19 (89.4%) of subjects deposited money in their deposit contracts and 14/17 participants who made initial deposits either held constant or increased their contributions each month. Subjects in both incentive groups lost significantly more weight on average than subjects in the control group (4.0 lbs) (lottery 13.1 lbs, p = 0.015; deposit contract 14.0 lbs, p = 0.003). Of the subjects not lost to follow-up in the two incentive arms (32 out of 38), all of them lost weight.

Based on this promising preliminary evidence and supplemental funding from the Hewlett Foundation, we propose an 8-month study with 2 intervention arms to further examine the effect of incentives on long term weight loss success. This study will build on the work to date to examine which intervention is most successful in promoting sustained weight loss. The proposed 3-arm extension will enroll 66 participants from Philadelphia VA with BMIs between 30 and 40, starting with those potential participants who were placed on a waiting list for our previous study after an overwhelming response to the initial mailing.

DETAILED DESCRIPTION:
The proposed study, a 3-arm randomized control trial (RCT), would be tested with 66 patients at Philadelphia VA with BMIs between 30 and 40. Participants in the control group would receive usual care from their providers and monthly weigh ins. Participants in the incentive conditions will receive daily monitoring of their weights for 32 weeks, plus a package of financial incentives if they lose weight. Incentive group subjects will be given a weight loss target of 24 lbs in the first 24 weeks and will be able to choose a weight loss goal of 0, 0.5, or 1 lb per week for the final two months of the study. Financial incentives in the first deposit contract condition will consist of a potential payment for every day they are under their target weight which consists of the prorated daily amount of their deposit contract plus an equal 1:1 match provided by the study team for the first 6 months framed as 'weight loss period' and then for 2 months framed as 'maintenance of weight loss'. In the second deposit condition, the incentive consists of 8 months of the prorated daily amount of their deposit contract plus a 1:1 match (without the framing of 'weight loss' vs 'maintenance of weight loss'). We will have 80% power to find a 5 kg difference in weight loss between the intervention and control groups. Subjects who lose more than 20 pounds in either of the intervention groups will be eligible for an additional incentive.

The proposed interventions will serve as the basis for a larger-scale intervention study of incentives for weight loss and maintenance that has the potential to substantially reduce the health burden of obesity among veterans.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30-40;
* Age between 30-70;
* At least moderately interested in losing weight (Self-reported 3,4, or 5 on 5 point scale)

Exclusion Criteria:

* Unstable medical conditions that would likely prevent the subject from completing the study;
* Myocardial infarction within 6 months;
* Uncontrolled hypertension, defined as BP>170 mm Hg systolic or BP>110 mm Hg diastolic;
* Diabetic using any medicine besides metformin to control blood sugars
* Metastatic cancer;
* Self-report of 6 or more alcoholic beverages per day;
* Severe depression;
* Active substance abuse;
* Schizophrenia
* Inability to read or severe cognitive deficits that would preclude ability to read consent form or fill out surveys).
* Participation in another research study unless copy of consent form obtained and screened for possible confounding of results.
* Those currently enrolled in a weight loss program elsewhere.
* Pregnant women

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
actual weight loss | eight months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD PhD, Principal Investigator — Philadelphia Veterans Administration Medical Center
Locations (1):
- Philadelphia Veterans Administration Medical Center, Philadelphia, Pennsylvania, United States